CLINICAL TRIAL: NCT04292665
Title: Randomized Controlled Trial of Classical Massage and Benson Relaxation Exercise for Patients With Heart Failure
Brief Title: Effects of Classical Massage and Benson Relaxation Exercise on Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Gulbahar, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure; Symptoms and Signs; Quality of Life
Keywords: Classical massage,heart failure,nursing,relaxation
MeSH Terms: conditions — Heart Failure; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classical Massage (Experimental): Patients will receive a total of fourteen individual applied classical massage sessions, twice daily for seven days, each session lasting 30 minutes.
  Interventions: Behavioral: Classical Massage
- Relaxation (Experimental): Patients will receive a total of fourteen individual counseling sessions, in a quiet room, twice daily for seven days, each session lasting 20 minutes.
  Interventions: Behavioral: Benson Relaxation Exercise
- Control (Other): Patients will continue to receive standard nursing care and no further intervention will be made during the research.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Classical Massage — During the first interview, a booklet explaining the introduction, purpose, benefits and application steps of hand-foot massage will be given to the patients in the classical massage group. Hand and foot massage will be applied to the patients for 30 minutes in the form of right hand five minutes, left hand five minutes, right foot ten minutes, left foot ten minutes, using liquid vaseline in each session twice a day in the patient's own bed with individual applied sessions by the researcher. Patients will receive a total of 14 sessions of classical massage, twice a day, for seven days.
  Arms: Classical Massage
Behavioral: Benson Relaxation Exercise — During the first interview, patients will be given a booklet explaining the description, purpose, benefits and application steps of the Benson relaxation exercise. With individual counseling sessions, a total of 14 sessions of Benson relaxation exercises will be performed in a quiet room, twice a day for seven days, each session lasting 20 minutes. At the beginning of the application, patients will focus on their breaths by taking slow and natural breaths with the researchers' commands and will quietly say to yourself the words of the focus, sound, sentence or prayer they choose, which are meaningful to them.
  Arms: Relaxation
Other: Control — Patients will continue to receive standard nursing care and no further intervention will be made during the research.
  Arms: Control

SUMMARY:
Patients with heart failure will be entered. Participants will be randomized to one of three study arms: Arm 1: Classical massage, Arm 2: Relaxation, Arm 3: Control Hypothesis: Classical Massage and Benson Muscle Relaxation will decrease frequency, severity, discomfort of symptoms and improve quality of life.

DETAILED DESCRIPTION:
Previous reports have revealed that classical massage and Benson relaxation exercise are promising for physiological parameters such as respiratory rate, pulse, blood pressure in heart failure patients. On the other hand, research examining effects of these approaches on physical symptom status that is including dyspnea, orthopnea, fatigue, chest pain, peripheral edema, sleep problems and dizziness and quality of life is limited. The present study investigates the effects of classical massage and Benson relaxation exercise in a single-site, 3-arm, randomized, controlled study of 96 patients with heart failure. Arm 1: Classical massage; Arm 2: Benson relaxation exercise; Arm 3: Control. The investigators hypothesize that Classical Massage and Benson relaxation exercise will decrease frequency, severity, discomfort of symptoms and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being at least primary school graduates,
* Being over 18 years old
* Being diagnosed Stage III-IV with heart failure
* Not using any other complementary or integrative therapy during the study period

Exclusion Criteria:

* Having an additional disease such as advanced stage chronic obstructive pulmonary disease, asthma, cancer
* Stage I-II diagnosed with heart failure
* Having an active thrombosis
* Having a coagulation problem
* Not volunteering to participate in the research
* Patients who have been hospitalized for 5 days or less and discharged before five days after the start of the application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in symptom status | Baseline measurements, at the end of 7th day and two weeks after the completion of the interventions
  Symptom status will be measured based on patient report by the Symptom Status Questionnaire-Heart Failure . Higher score means increase in symptom burden.
Change in quality of life | Baseline measurements, at the end of 7th day and two weeks after the completion of the interventions
  Quality of live will be measured by the Minnesota Living with Heart Failure Questionnaire. Higher scores on the scale mean worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Gok Metın, Assos.Prof., Study Director — Hacettepe University
Locations (1):
- Ankara University Medical Faculty Ibni Sina Hospital Cardiology Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No